CLINICAL TRIAL: NCT02568891
Title: Modulation of Gut Microbiota in End-stage Renal Disease: A Pilot Study
Brief Title: Modulation of Gut Microbiota in End-stage Renal Disease
Acronym: MGM-dialysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding obtained
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 26-255 ex 13/14
Record Dates: First submitted 2015-07-29; First posted 2015-10-06 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): 6 g of Winclove-849 containing Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus salivarius W24, Lactococcus lactis W19, Lactococcus lactis W58 at a concentration of 2.5 x 109 cfu/g
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): similar looking and tasting placebo without bacteria
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — multispecies probiotic
  Arms: Probiotic
Dietary Supplement: Placebo — matrix
  Arms: Placebo

SUMMARY:
In end-stage renal disease (ESRD) cardiovascular and infectious complications are common. The gut microbiome might play an important pathophysiological role. ESRD is hypothesized to be associated with profound alterations of gut microbiome and gut permeability. The investigators aim to test whether a multispecies probiotic mixture is able to revert the microbiome changes and decrease gut permeability. Furthermore the investigators aim to test whether this improvement in microbiome composition and gut permeability is also associated with improvements in endotoxemia, uremia and cardiovascular risk factors.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) has a prevalence of 10% in the general population and up to 20% in high-risk groups, such as patients with diabetes. Despite the widespread availability of renal replacement therapy in the western world, mortality of patients with end-stage renal disease (ESRD) is still high. The life expectancy of patients with renal replacement therapy in Austria is reduced by more than 50%.

Patients on renal replacement therapy exhibit an increased cardiovascular mortality (10-30 fold higher than in the general population) associated with accelerated vascular calcification. The KIDNEY DISEASE IMPROVING GLOBAL OUTCOMES (KDIGO)-work group introduced the term CKD-Mineral and Bone Disorder (CKD-MBD) which describes a clinical syndrome encompassing mineral, bone, and calcific cardio-vascular abnormalities that develop as a complication of CKD. This syndrome emerges as a result of a declining kidney function and is characterized by changes of circulating levels of parathyroid hormone (PTH), 25-hydroxyvitamin D (25(OH)D),1,25-dihydroxyvitamin D (1,25(OH)2D), other vitamin D metabolites and fibroblast growth factor-23 (FGF-23). The ability of the failing kidneys to excrete phosphate is diminished and hyperphosphatemia occurs. High phosphate levels together with calcium as well as low concentrations of fetuin A, the main calcification inhibitor under physiological conditions, lead to increased vascular and extravascular calcification and renal bone disease. Another important calcification inhibitor is the vitamin K2-dependent matrix Gla-protein (MGP). Dialysis patients exhibit a low vitamin K intake and suffer substantially from vitamin K deficiency. Insufficient vitamin K intake leads to the production of non-carboxylated, inactive MGP and deficiency of carboxylated MGP may contribute substantially to the development and progression of arterial calcification. Bacterial infection and sepsis, although decreasing over the last decades, also account for up to 20% of deaths in ESRD-patients and are the second most common cause of mortality and hospitalization. Mortality due to sepsis is 100 - 300 times higher in dialysis patients as compared to the general population. The mechanisms of the increased susceptibility to infection are unclear but recent studies suggest that in patients with ESRD, innate immune response is defective. One reason for defective innate immunity might lie in an increased risk for endotoxemia. Hemodialysis (HD)-induced regional splanchnic ischemia leads to increased gut permeability and consecutive endotoxin translocation. This possibly results in alterations in gut microbiome composition.

Recently profound alterations of the composition of the gut microbiome in ESRD have been shown. In ESRD subjects, more Firmicutes, Actinobacteria and Proteobacteria and fewer Sutterellaceae, Bacteroidaceae, and Lactobacillaceae were observed relative to controls. The frequent use of antibiotics, phosphate binders and an often polypragmatic drug consumption has a considerable impact on the microbiome of ESRD-patients.

These alterations of gut microbiota can impact on several mechanisms in ESRD. Gut bacteria produce vitamin K and the microbiome composition might therefore play a pivotal role in providing enough vitamin K for a sufficient carboxylation of MGP, a potent inhibitor of arterial calcification. Treatment with vitamin K antagonists, for example, has been associated with a 10 fold increased risk for the development of calcification and calciphylaxis, a life threatening calcifying arteriolopathy in CKD-patients. Furthermore the gut is a potential source of endotoxin in patients with ESRD, due to translocation of bacterial products across the gastrointestinal barrier. In ESRD the presence of endotoxin is an independent predictor for mortality. Ultrafiltration during hemodialysis treatment leads to critical ischemia in the splanchnic vascular bed, thus adversely affecting the integrity of the gut barrier. Disruption of gut barrier function in ESRD allows translocation of endotoxin and bacterial metabolites to the systemic circulation, which contributes to inflammation and uremia and prompts progression of the disease. Furthermore, subclinical inflammation in ESRD-patients has been shown to promote progression of cardiovascular disease as well. The gut microbiome also impacts on glucose metabolism and plays a critical role in obesity and the development of insulin resistance and type 2 diabetes. Protein fermentation by gut microbiota generates toxic metabolites and many of the known uremic toxins are of intestinal origin, including p-cresol and indoxyl sulfate. Modulation of the microbiome can contribute to the reduction/elimination of uremic toxins.

Improving the poor prognosis of ESRD patients is an ongoing challenge. An increased awareness of the limitations in conventional dialysis techniques has renewed interest in alternative therapeutics in recent years. An unmet clinical need for adjuvant therapeutic strategies persists in patients whether renal transplantation is intended or not. Supplementation of probiotics and thereby targeting the intestine, an important source of endotoxin and uremic toxins, might be a promising approach to partly overcome the high morbidity and mortality in ESRD patients. Probiotics are living beneficial microorganisms, able to gastroduodenal passage and maintain viability throughout the gut. Feasibility of gut microbiome modulation in ESRD was shown in animal and human settings. However, so far, it is unknown to what extend probiotics are able to re-establish gut microbiome homeostasis in ESRD. Furthermore the effects of a probiotic intervention on cardiovascular risk factors, inflammation, gut barrier and uremia have not been studied in detail yet.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patients with end-stage renal disease [5] undergoing any modality of renal replacement therapy (hemodialysis, hemodiafiltration or peritoneal dialysis)

Exclusion Criteria:

* Malignancy
* Pregnancy
* Chronic inflammatory bowel disease
* Celiac disease
* Active alcohol abuse (>40g alcohol per day)
* Any severe organ dysfunction unrelated to renal dysfunction

  20 healthy family members (living in the same household) of patients will be recruited as controls

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome | 1 year
  changes in gut microbiome composition

SECONDARY OUTCOMES:
gut permeability (zonulin in stool) | 1 year
  changes in gut permeability
bacterial translocation (bacterial DNA in serum) | 1 year
  decrease in bacterial translocation
neutrophil phagocytic capacity | 1 year
  improvement in neutrophil function
glucose metabolism (meal tolerance test) | 1 year
  improvement in glucose metabolism
uremia toxins | 1 year
  decrease in uremia toxins

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer, MD, Principal Investigator — Medical University of Graz; Harald Sourij, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria